CLINICAL TRIAL: NCT00122876
Title: A Phase 1/2 Open-Label Study to Evaluate Safety and Preliminary Evidence of Effectiveness of Tumor Ablation With Talaporfin Sodium (LS11) and Interstitial Light Emitting Diodes (LEDs) in the Treatment of Subjects With Inoperable Hepatocellular Carcinoma (HCC)
Brief Title: Tumor Ablation With Talaporfin Sodium and Interstitial Light Emitting Diodes Treating Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Organization: Light Sciences LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSC-OL004
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms
Keywords: Hepatocellular Carcinoma; HCC; Photodynamic therapy; Talaporfin Sodium (LS11); Light emitting diodes (LEDs); Litx; Light Infusion Technology
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Photochemotherapy; Talaporfin

INTERVENTIONS:
Procedure: Photodynamic therapy
Drug: Talaporfin Sodium

SUMMARY:
The purpose of this study is to determine whether the Litx™ treatment is safe and effective in treating inoperable hepatocellular carcinoma (HCC).

Litx™ is an integrated treatment system comprising an intravenously administered photosensitizing agent, Talaporfin Sodium (LS11), that is activated by non-coherent light generated inside the tumor by an implanted light emitting diode (LED) array light source.

DETAILED DESCRIPTION:
Subjects that provide Informed Consent and satisfy the Eligibility Criteria will undergo CT or Ultrasound guided percutaneous placement of a single, two, three, or four Light Sources depending on their tumor characteristics. No more than four Light Sources will be used at a single treatment session. The Light Sources may be used in a single lesion or in multiple lesions. Depending on lesion size, one or more Light Sources may be used to treat a single lesion.

Following ultrasound or CT confirmation of the Light Sources, patients will receive an intravenous dose of LS11 at 1 mg/kg. 15 minutes to 1 hour following completion of LS11 administration, delivery of 200 J/cm light energy at 20 mW/cm will begin. Upon completion of light treatment, the Light Sources will then be manually removed and the patients will be observed for acute complications.

Subjects will be evaluated for treatment-related adverse events at every scheduled clinical visit. Restaging by contrast enhanced spiral CT and tumor evaluation, using the RECIST criteria, are performed at Week 4 and Week 8.

Subjects may receive a second Litx™ treatment at Week 4 or Week 8, as recommended by the study investigator. Subjects who receive the second Litx™ treatment will be evaluated for treatment-related adverse events at every scheduled clinical visit. Restaging by contrast enhanced spiral CT and tumor evaluation, using the RECIST criteria, are performed. The active phase of the protocol ends 8 weeks after the last treatment received.

Following completion of the active phase of the protocol, subjects will be monitored for survival for one year (at 6, 9 and 12 month time points) from the date of study entry or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary Hepatocellular Carcinoma (HCC), established by any one of the following criteria in a clinical setting suggestive of HCC: (i) Two different imaging techniques that suggests HCC; (ii) Combination of one imaging technique that suggests HCC and serum alpha-fetoprotein (AFP) level >400 ng/mL; (iii) Histological evidence of HCC;
* Subjects with at least 1 but no more than 3 lesions in the liver may be considered for enrollment in the study;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* Life expectancy of at least 16 weeks;
* Prior treatment failure with locally ablative techniques is allowed. Subjects who were not candidates for surgery, systemic chemotherapy, chemoembolization (TACE), intratumoral ethanol injection (PEI), radiofrequency ablation (RFA), cryoablation or other locally ablative technology may be eligible, but at least 4 weeks must have elapsed since the completion of any prior therapy and the subject must have recovered from acute side effects;
* Understanding and ability to sign written informed consent;
* 18 years of age or more;
* Adequate hematologic, liver and renal functions as evidenced by the following: *WBC > 2,400/mm; *Platelet Count > 75,000/µl; *Hemoglobin > 9.4 gm/dL; *PT and PTT < 1.5 Control; *AST, ALT < 5 x ULN; *Bilirubin < 1.5 X ULN; *Alk Phos < 3X ULN; *Creatinine < 2.5 mg/dL (SI: 221 mmol/L)

Exclusion Criteria:

* Subjects who are candidates for surgery with curative intent;
* Subjects with lesions larger than 8 cm in diameter and more than 40% of parenchymal disease involvement;
* Known sensitivity to porphyrin type drugs;
* Known history of porphyria;
* Known presence of extrahepatic metastases;
* Anticipated need for systemic chemotherapy during the first 8 weeks of the study;
* Child-Pugh C cirrhosis;
* Diffuse HCC;
* Concurrent participation in another clinical trial involving experimental treatment;
* Any concurrent disease or condition that in the opinion of the investigator impairs the subject's ability to complete the trial. Psychological, familial, sociological, geographical or medical conditions which in the Principal Investigator's opinion could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial's data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Tumor Response
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Sy-Shi Wang, PhD, Study Director — Light Sciences Oncology
Locations (9):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore
- Taiwan (6):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung Hsien
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan Hsien

REFERENCES:
- [Background] Lustig RA, Vogl TJ, Fromm D, Cuenca R, Alex Hsi R, D'Cruz AK, Krajina Z, Turic M, Singhal A, Chen JC. A multicenter Phase I safety study of intratumoral photoactivation of talaporfin sodium in patients with refractory solid tumors. Cancer. 2003 Oct 15;98(8):1767-71. doi: 10.1002/cncr.11708. PMID 14534895
- [Background] Chen J, Keltner L, Christophersen J, Zheng F, Krouse M, Singhal A, Wang SS. New technology for deep light distribution in tissue for phototherapy. Cancer J. 2002 Mar-Apr;8(2):154-63. doi: 10.1097/00130404-200203000-00009. PMID 11999949